CLINICAL TRIAL: NCT04045587
Title: International Severe Asthma Registry: Canadian Cohort
Acronym: ISAR
Status: Recruiting | Type: Observational
Sponsor: University of British Columbia (Other)
Collaborators: University of Alberta (Other); University of Toronto (Other); Laval University (Other); McGill University (Other); Université de Sherbrooke (Other); The Ottawa Hospital (Other); Queen's University (Other); University of Saskatchewan (Other); Western University, Canada (Other)
Responsible Party: Principal Investigator, Celine Bergeron, Principal Investigator, University of British Columbia
Other Study IDs: H17 - 03052
Record Dates: First submitted 2019-07-31; First posted 2019-08-05 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Severe Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Severe Asthma Participants: Participants with severe asthma classified at GINA Step 4 and uncontrolled in terms of their symptoms and exacerbations or GINA Step 5.

SUMMARY:
The International Severe Asthma Registry is a global initiative looking to ensure that the care of people with severe asthma will continue to improve by collecting detailed information about the health and treatment of as many people with the disease as possible. The study will gather anonymized longitudinal real-life data for participants with severe asthma for five years. The purpose of the registry is to track the progress of participants and determine how well they are responding to treatment. Medical research using data from the registry will give the investigators a better understanding of severe asthma and help the investigators develop and improve the care and treatment for severe asthma participants. The Canadian cohort of the registry will collect information from Canadian participants with severe asthma across seven different sites.

DETAILED DESCRIPTION:
Study staff will collect medical information through reviewing participant medical charts and interviewing participants about their health/asthma. The information collected includes birth date, gender, ethnicity, height/weight, body mass index, medical history (smoking history and exacerbation history), current and past asthma related medications, and any recent test results available pertaining to blood work, lung function, allergen skin prick, and imaging. This information will be collected at the baseline visit, and then once a year at a follow up visit, for five years (total of five visits).

Participants will be assigned a unique study number to protect the confidentiality of their personal health care information. All study data will be de-identified and then stored in a secure information management system, hosted at the study sponsor, Optimum Patient Care Global Limited in Cambridge, United Kingdom. Participant identities will always be kept confidential and will not be included in any research that is published. Data collected across the Canadian sites will be used to find ways to improve asthma treatments in Canada, to report on current patterns of managing severe asthma in Canada, to identify different sub-groups of severe asthma, and to carry out various medical research to understand asthma better and develop new treatments.

Research records and health or other source records may be inspected in the presence of the Principal Investigator or by representatives of the University of British Columbia's Clinical Research Ethics Board for the purpose of monitoring the research. No information or records that disclose participants' identities will be published without subject consent, nor will any information or records that disclose participants' identities be removed or released without subject consent unless required by law.

ELIGIBILITY:
Inclusion Criteria:

* Participants 18 years or older
* Participants receiving treatment according to GINA Step 5 or uncontrolled in GINA Step 4 (uncontrolled is defined as having severe asthma symptoms or frequent exacerbations)

Exclusion Criteria:

-Participants with mild to moderate asthma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be selected from respirology/pulmonary clinics across Canada. Participants will be identified and recruited by the study investigators and study staff based on their clinical presentation.
Sampling Method: Non-Probability Sample
Enrollment: 714 (Estimated)
Dates: Start 2018-11-06 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Blood eosinophil counts | Past 12 months
  10^9/L
Blood Immunoglobulin E (IgE) counts | Past 12 months
  kilo unit/L
Fractional exhaled nitric oxide level | Past 12 months
  parts per billion
Start and end dates of oral corticosteroid medication | Prior to baseline visit
  Day/Month/Year for start and end dates if available
Asthma Control | Past 4 weeks
  Assessed through the Global Initiative for Asthma (GINA) Questionnaire
Start and end dates of biologic medications such as anti-interleukin-5, anti-immunoglobulin E, or anti-interleukin-4 treatments (if relevant) | Prior to baseline visit
  Day/Month/Year for start and end dates if available
Reason for switching biologic medication (if relevant) | Past 12 months
  Options include: lack of clinical efficacy, side effects, biologic access restriction, and patient preference
Start and end dates of all asthma related inhaled medications | Prior to baseline visit
  Day/Month/Year for start and end dates if available
Number of asthma exacerbations requiring rescue steroids | Past 12 months
  Severe asthma exacerbations are defined as events that require urgent action (rescue steroids) by the participant and physician to prevent a serious outcome
Number of emergency room visits for asthma | Past 12 months
  Total number of visits
Number of hospital admissions for asthma | Past 12 months
  Total number of admissions
Spirometry test results for Forced Vital Capacity (FVC) | Past 12 months
  Pre- and post-bronchodilator FVC results in litres
Spirometry test results for Forced Expiratory Volume in One Second (FEV1) | Past 12 months
  Pre- and post-bronchodilator FEV1 results in litres

CONTACTS AND LOCATIONS:
Overall Officials: Celine Bergeron, Principal Investigator — University of British Columbia
Locations (11):
- Canada (11):
  - University of Alberta, Edmonton, Alberta
  - Synergy MD Specialty Group, Edmonton, Alberta
  - University of British Columbia, Vancouver, British Columbia
  - Kingston General Hospital, Kingston, Ontario
  - University of Western Ontario, London, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - Inspiration Research Limited, Toronto, Ontario
  - McGill University, Montreal, Quebec
  - Université de Sherbrooke, Sherbrooke, Quebec
  - Université Laval, Quebéc City, Quebéc
  - University of Saskatchewan, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: No